CLINICAL TRIAL: NCT03984591
Title: Cluster and Registry Trials Of the Working Group of Heart Failure in Denmark: Are SPironolactone and Eplerenone Comparable Treatments?
Brief Title: A Registry-based Cluster Randomized Trial to Compare the Effect of Spironolactone vs. Eplerenone on Clinical Outcomes in Patients With Symptomatic Systolic Heart Failure
Acronym: CROWD-ASPECT
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Jakob Thune, Clinical research associate professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROWD-ASPECT
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Systolic Heart Failure
Keywords: aldosterone antagonists; spironolactone; eplerenone; mortality
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Eplerenone; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Active Comparator): Spironolactone used according to heart failure guidelines
  Interventions: Drug: Spironolactone
- Eplerenone (Active Comparator): Eplerenone used according to heart failure guidelines
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Eplerenone according to guidelines
  Arms: Eplerenone
Drug: Spironolactone — Spironolactone according to guidelines
  Arms: Spironolactone

SUMMARY:
Objective The objective is to compare the efficacy of spironolactone and eplerenone on clinical outcome in patients with heart failure and a reduced ejection fraction.

Method The study is a crossover cluster randomized trial. Each heart failure clinic in Denmark will be allocated to four periods (clusters): two periods with spironolactone and two periods with eplerenone as first drug. The planned total participation time for each department is 4 years and we estimate that data from 7200 patients will be accrued in this period. Endpoints will be assessed through Danish National Registries.

ELIGIBILITY:
Inclusion Criteria:

* all patients registered in the Danish Heart Failure Registry who has a baseline left ventricular ejection fraction <40% and who has filled in a prescription for an aldosterone antagonist

Exclusion Criteria:

* patients who had filled in a prescription for an aldosterone antagonist prior ro registration in the Danish Heart Failure Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Mortality (will be used if overall mortality rate is 15% or greater)
Mortality or hospitalization for heart failure | 6 years
  Will be used if overall mortality is less than 15%

CONTACTS AND LOCATIONS:
Overall Officials: Jens Jakob Thune, MD, PhD, Study Chair — Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data is located on research servers with Statistics Denmark. Individual participant data may not be exported from the servers.